CLINICAL TRIAL: NCT03998202
Title: Myopenia and Mechanisms of Chemotherapy Toxicity in Older Adults With Colorectal Cancer: The M&M Study
Brief Title: Myopenia and Mechanisms of Chemotherapy Toxicity in Older Adults With Colorectal Cancer
Acronym: M&M
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00058811; NCI-2019-02514 (Registry Identifier: NCI Trial Identifier [CTRP]); WF-1806 (Registry Identifier: LPO ID); IRB00058811 (Other: WF eIRB ID)
Record Dates: First submitted 2019-06-21; First posted 2019-06-26 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer; Sarcopenia
Keywords: Colorectal Cancer; Myopenia; Sarcopenia; Chemotherapy; Geriatric-Oncology
MeSH Terms: conditions — Colorectal Neoplasms; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood obtained for DNA extraction
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adults 60-74 years
- Adults >= 75 years

SUMMARY:
This study will examine the association between low muscle mass (myopenia) at diagnosis and chemotherapy toxicity in older adults with newly diagnosed advanced colorectal cancer.

DETAILED DESCRIPTION:
This is a prospective cohort study that examines the impact of myopenia on chemotherapy toxicity in overall survival (OS) in older adults with newly diagnosed metastatic colorectal cancer (CRC) receiving 5-Fluouracil (5FU)systemic chemotherapy. The study also explores the mediating influence of genetic variation in the association between myopenia and chemotherapy toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed metastatic CRC or newly recognized metastatic recurrence of CRC >= to 3 months (12 weeks) from completion of treatment of non-metastatic CRC.
* Planning to or recently started to undergo undergo immunotherapy and/or 5-FU based chemotherapy as a first line of treatment. 5-FU chemotherapy can be 5-FU alone or in combination with oxaliplatin and/or irinotecan +/- immunotherapy. Capecitabine is also acceptable.
* Estimated life expectancy >= 6 months.
* Patients must be able to comprehend English or Spanish (for questionnaire completion).
* Ability to understand and the willingness to sign a written informed consent document.
* Patient eligibility is not dependent on BMI or weight. Patients with a significant (+- > 10%) body weight change in the previous 12 months are eligible for this study.

Exclusion Criteria:

* Patients enrolled on hospice.
* Prior systemic chemotherapy for metastatic colorectal cancer (ok if adjuvant chemotherapy completed >= 3 months (12 weeks) prior to this disease disease recurrence and treatment).
* Patients may not be receiving any other investigational agents.
* No untreated brain metastases. Patients with treated brain metastases are eligible.
* Patients on or planned to undergo radiation therapy in near future.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed metastatic CRC or metastatic recurrence of CRC >= 3 months (12 weeks) from diagnosis at 60 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-09-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Chemotherapy Toxicities (Grade 3 - 5) | Up to 6 months (after initiation of chemotherapy)
  Chemotoxicity will be measured after initiation of chemotherapy using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE).

SECONDARY OUTCOMES:
Overall Survival | 1 year
  Participants will be followed for the duration of the study with each participant followed for at least one year after diagnosis, to determine vital status. Loss-to-follow-up will be minimized by asking participating sites to provide date of last contact every 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Lesser, MD, Study Chair — WFUSM
Locations (146):
- United States (146):
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - John B Amos Cancer Center, Columbus, Georgia
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Carle Physician Group - Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - The University of Iowa - Ankeny, Ankeny, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - The University of Iowa-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - MBP Cancer Center - Baton Rouge General, Baton Rouge, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology-Brighton, Brighton, Michigan
  - Trinity Health Medical Center-Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Hematology Oncology Consultants-Chelsea Hospital, Chelsea, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Marshfield Medical Center Dickinson, Iron Mountain, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology -Ann Arbor, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Levine Cancer Institute-SouthPark, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Levine Cancer Institute-Gaston, Gastonia, North Carolina
  - Wake Forest Baptist Health - Wilkes Medical Center, Wilkesboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Adena Regional Medical Center, Chillicothe, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Wake Forest NCORP Research Base is committed to following the NIH Statement on Sharing Research Data (http://grants.nih.gov/grants/guide/notice-files/NOT-OD-03-032.html). As of July 2018, the WF NCORP RB signed an agreement with NCI to contribute de-identified data and data dictionaries from clinical trials conducted through our RB to the NCI NCTN/NCORP data archive within 6 months of primary and non-primary publications of phase II/III and phase III trials to https://nctn-data-archive.nci.nih.gov/. This will become the primary means for sharing raw data, and we will adhere to the guidelines spelled out in the NCTN/NCORP Data Archive Usage Guide. De-identified data from studies not covered by the agreement (e.g., phase II and observational studies) will be made available upon request. All data files will be de-identified. De-identification procedures will meet the HIPAA criteria as detailed in the Code of Federal Regulations, Part 45, Section 164.514.
Time Frame: 6 months after publication for a 2 year duration
Access Criteria: upon to request to NCORP@wakehealth.edu